CLINICAL TRIAL: NCT06883396
Title: JUPITER 4.0 - Risk Factors for Failure of Isolated Medial Patellofemoral Ligament Reconstruction
Status: Recruiting | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: American Orthopaedic Society for Sports Medicine (Other); Orthopedic Research and Education Foundation (Other); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-0649
Record Dates: First submitted 2025-01-22; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-01

CONDITIONS: Patellar Dislocation, Recurrent; Patellar Dislocation; Patellar Instability; Patellofemoral Dislocation; Patellofemoral Joint Dislocation; Patellofemoral Disorder
Keywords: Patella; Patella Dislocation; Patellar Instability; Recurrent Patellar Instability; MPFL; Medial Patellofemoral Ligament; Medial Patellofemoral Ligament Reconstruction; Patellofemoral Instability
MeSH Terms: conditions — Patellar Dislocation; Recurrence; Patella Fracture | interventions — Plastic Surgery Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Isolated MPFL Reconstruction: Patients with recurrent patellar instability (2 or more dislocation and/or subluxation events) undergoing isolated MPFL reconstruction
  Interventions: Procedure: Medial Patellofemoral Ligament (MPFL) Reconstruction

INTERVENTIONS:
Procedure: Medial Patellofemoral Ligament (MPFL) Reconstruction — For the purposes of this study, isolated MPFL reconstruction is defined as MPFL reconstruction with a tendon graft, with or without additional soft tissue procedure(s) including lateral retinacular lengthening or release, patellofemoral chondroplasty and/or cartilage restoration. No patient in the study will receive a bony realignment procedure to treat patellar instability.

SUMMARY:
The goal of this observational study is to learn about the outcomes of medial patellofemoral ligament (MPFL) reconstruction for the treatment of recurrent patellar instability. The main questions it aims to answer are:

* What are the risk factors for recurrent patellar instability after MPFL reconstruction?
* What functional outcomes do patients report after MPFL reconstruction?

Participants undergoing MPFL reconstruction will answer survey questions about their knee and activity level 1 year and 2 years after surgery.

DETAILED DESCRIPTION:
The JUPITER group consists of high-volume patellofemoral surgeons across the United States, and was organized to facilitate the collection of clinical and radiographic outcomes following surgical and non-surgical treatment of patellar instability. With this study (JUPITER 4.0), the group aims to prospectively enroll a new cohort of consecutive patients with recurrent patellar instability that would undergo isolated MPFL reconstruction regardless of radiographic measurements or anatomic risk factors to address two specific aims - 1) what patient, injury, and surgical factors lead to recurrent instability following isolated MPFL reconstruction and 2) the creation of an instability severity index score, with the long-term objective of identifying preoperatively, patients with a high risk of failure of an isolated MPFL reconstruction who may be better served with concomitant bony procedure.

ELIGIBILITY:
Inclusion Criteria:

* 10-35 years old
* Recurrent patellar instability with at least one episode defined as either (1) a dislocated patella requiring reduction in the emergency department or (2) a convincing history for dislocation, associated with full giving way, and the following physical findings: (a) hemarthrosis or effusion, (b) tenderness along the medial retinaculum, and (c) apprehension when laterally directed force was applied to the patella or (3) MRI-documented dislocation with associated bone bruises

Exclusion Criteria:

* Previous ipsilateral knee surgery
* Obligatory/fixed/habitual patella dislocation or subluxation
* Unloadable inferior or lateral chondral damage on the patella that would require a tibial tubercle transfer for unloading purposes
* Pathologic tibiofemoral instability

Ages: 10 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients presenting to the participating surgeons for treatment of recurrent patellar instability
Sampling Method: Non-Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Recurrent patellar instability | Within 24 months post-operatively
  Patient-reported patellar dislocation or subluxation

SECONDARY OUTCOMES:
Patient-Reported Outcome Measures (PROMs): Kujala score | 12 months post-operatively and 24 months post-operatively
  The Kujala score, also known as the Anterior Knee Pain Scale (AKPS), is a 13-item questionnaire that helps assess subjective reactions to activities and symptoms related to patellofemoral pain. It is a 0-to-100 point scale, with higher scores indicating better outcomes and less pain and disability.
Patient-Reported Outcome Measures (PROMs): Pedi-IKDC | 12 months post-operatively and 24 months post-operatively
  The Pedi-IDKC is a modified version of the International Knee Documentation Committee (IDKC) Subjective Knee Form for use in young patients. It is a 15-item knee-specific questionnaire that measures symptoms, function, and sports activity. Scores range from 0-100, with higher scores indicating better outcomes.
Patient-Reported Outcome Measures (PROMs): HSS Pedi-FABS | 12 months post-operatively and 24 months post-operatively
  The Hospital for Special Surgery Pediatric Functional Activity Brief Scale (HSS Pedi-FABS) is a validated 8-item questionnaire scored from 0-30, with higher scores indicating higher levels of activity.
Patient-Reported Outcome Measures (PROMs): KOOS-12 | Time Frame: 12 months post-operatively and 24 months post-operatively
  The Knee injury and Osteoarthritis Outcome Score-12 (KOOS-12) is a 12-item measure evaluating the difficulties people experience due to problems with their knee. Each question is scored from 0 to 4 points, with 0 representing no knee problems and 4 representing extreme knee problems. Overall, scores range from 0 to 100, where, in contrast to the individual questions, 0 is the worst possible and 100 is the best possible score.
Patient-Reported Outcome Measures (PROMs): BPII 2.0 | 12 months post-operatively and 24 months post-operatively
  The BPII 2.0 (Banff Patellofemoral Instability Instrument) is a patient-reported outcome measure assessing quality of life in individuals with patellofemoral instability. The score ranges from 0 to 100, with higher scores indicating greater quality of life.
Patient-Reported Outcome Measures (PROMs): PROMIS-29 | 12 months post-operatively and 24 months post-operatively
  PROMIS (Patient-Reported Outcomes Measurement Information System) is a questionnaire that evaluates health-related quality of life across seven key domains: physical function, pain interference, fatigue, sleep disturbance, physical and mental health, and social health. It is scored a T-score metric. High scores mean more of the concept being measured. 10 points on the T-score metric is one standard deviation (SD).

CONTACTS AND LOCATIONS:
Overall Officials: Beth Shubin Stein, MD, Principal Investigator — Hospital for Special Surgery, New York; Shital Parikh, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (16):
- United States (16):
  - Stanford University, Redwood City, California
  - University of Florida, Gainesville, Florida
  - Midwest Orthopaedics at Rush, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Mount Sinai, New York, New York
  - NYU Langone Health, New York, New York
  - Hospital for Special Surgery, New York, New York
  - Duke Health, Wake Forest, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Wexler Medical Center, Dublin, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Scottish Rite for Children, Dallas, Texas